CLINICAL TRIAL: NCT06157866
Title: Cognitive Training to Enhance Brain-to-brain Concordance During Acupuncture
Brief Title: Cognitive Training to Enhance Brain Concordance During Acupuncture
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Spaulding Rehabilitation Hospital (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Vitaly Napadow, LICAC, PhD, Professor, Spaulding Rehabilitation Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 2023P003155
Record Dates: First submitted 2023-11-05; First posted 2023-12-06 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Fibromyalgia
Keywords: hyperscan fmri; hyperscan EEG; acupuncture; fibromyalgia; chronic pain
MeSH Terms: conditions — Fibromyalgia; Chronic Pain | interventions — Electroacupuncture; Cognitive Training; Sex Education

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Training (Experimental): Participants will meet with a pain specialist who will conduct a specific form of cognitive training targeting fibromyalgia.
  Interventions: Other: Electroacupuncture; Behavioral: Cognitive Training
- Education Training (Active Comparator): Participants will meet with a pain specialist to receive education training related to fibromyalgia.
  Interventions: Other: Electroacupuncture; Behavioral: Education Training

INTERVENTIONS:
Other: Electroacupuncture — During the treatment sessions the acupuncturist will insert needles in several locations aimed to reduce the patient's fibromyalgia pain. A low-amplitude, sub-sensory electrical current will be activated by the acupuncturist.
Behavioral: Cognitive Training — Cognitive training with a pain specialist.
  Arms: Cognitive Training
Behavioral: Education Training — Education training with a pain specialist.
  Arms: Education Training

SUMMARY:
This study will evaluate the impact of a novel non-pharmacological multimodal therapy, a type of approach known to improve pain outcomes and recommended by the Institute of Medicine report for chronic pain management. This study design will also allow the investigators to evaluate a neural model supporting therapeutic alliance for pain outcomes for fibromyalgia.

DETAILED DESCRIPTION:
The patient-clinician interaction is central to most therapies and is supported by key interpersonal mechanisms of action such as clinician empathy, therapeutic alliance, and trust. However, the neural underpinnings of this effect are mostly unknown. The investigators' recently published study applied functional MRI (fMRI) hyperscanning (i.e. simultaneously neuroimaging chronic pain patients and clinicians in synchronized MRI scanners) demonstrated that brain-to-brain concordance in the temporoparietal junction (TPJ) is up-regulated following a clinical interaction and associated with patient analgesia. Fibromyalgia is a chronic pain disorder in great need of novel therapies. This study will evaluate the impact of a novel multimodal therapy, a type of approach known to improve pain outcomes and recommended by the Institute of Medicine report for chronic pain management. The study design will also allow the investigators to evaluate a neural model supporting therapeutic alliance for pain outcomes for fibromyalgia wherein training and acupuncture will synergistically target a critical therapeutic pathway - i.e., patient-provider alliance, instantiated by TPJ concordance.

ELIGIBILITY:
Inclusion Criteria:

* Meet traditional American College of Rheumatology (ACR) criteria for FM as well as the more recent Wolfe et al 2011 criteria
* Are on stable doses of medication for 30 days prior to entering the study and agree not to change medications or dosages during the trial
* Ability to fully understand and consent to study procedures
* Baseline pain intensity of at least 4/10
* Pain duration of at least 6 months

Exclusion Criteria:

* Any longer period of work experience involving pain treatment, pain rehabilitation etc.
* Presence of any illness that is judged to interfere with the trial. For example: psychiatric disorder according to the DSM-IV manual
* Presence of any contraindications to fMRI scanning. For example: cardiac pacemaker, metal implants, fear of closed spaces, pregnancy.
* History of significant head injury
* Inability to respond accurately to the pain-relieving intervention in the behavioral part of the experiment, indicating a lack of response to the expectancy manipulation. If the healthy volunteer or clinician is not a responder to the behavioral expectancy induction he or she will be excluded.
* Unwillingness to receive brief experimental pain.
* Leg pain or health issues that may interfere with the study procedures.
* Comorbid acute pain condition
* Comorbid chronic pain condition that is rated by the subject as more painful than fibromyalgia
* Current use of opioid analgesics
* Concurrent inflammatory or autoimmune disease
* Documented peripheral neuropathy
* Pregnant
* Any psychiatric disorder involving a history of psychosis (e. g schizophrenia, bipolar disorder, severe personality disorders)
* History of anxiety disorders or significant anxiety symptoms interfering with fMRI procedures (e.g., panic)
* Psychiatric hospitalization in the past 6 months
* Unwillingness to withhold from consuming marijuana 12 hours prior to scans
* Unwillingness to withhold from consuming nicotine 4 hours prior to scans
* Any impairment, activity or situation that in the judgment of the Study Coordinator or Principal Investigator would prevent satisfactory completion of the study protocol.
* Is an actual clinical patient of the clinician subject
* Recent history of formal meditation-based training

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-02-16 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Brain Imaging-fMRI | Up to 6 months
  Hyperscan fMRI assessing brain-to-brain concordance between the patient and the clinician.

SECONDARY OUTCOMES:
Brain Imaging-EEG | Up to 6 months
  Hyperscan EEG assessing brain-to-brain concordance between the patient and the clinician.

OTHER OUTCOMES:
Brief Pain Inventory (BPI) - Pain Interference | Up to 6 months
  Brief Pain Inventory (BPI) is a validated 16 item questionnaire designed to assess the severity and interference of pain experienced. Pain interference is assessed on a scale from 0 (no interference) to 10 (severe interference).

CONTACTS AND LOCATIONS:
Overall Officials: Vitaly Napadow, PhD, Principal Investigator — Spaulding Rehabilitation Hospital
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Charlestown, Massachusetts
  - Spaulding Rehabilitation Hospital, Charlestown, Massachusetts
  - Brigham and Women's Hospital, Chestnut Hill, Massachusetts

IPD SHARING:
Plan to Share IPD: No
Per NIH guidelines